CLINICAL TRIAL: NCT02763098
Title: Effects of Different Doses of Remifentanil on Hemodynamic Response to Anesthesia Induction in Elderly Patients
Brief Title: Remifentanil on Hemodynamic Response to Anesthesia Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Nilay Boztas,MD, MD, Consultant, Dept of Anesthesiology and Reanimation, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 2012/25-04
Record Dates: First submitted 2016-04-13; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Anesthesia
Keywords: cardiovascular responses; analgesics opioid; remifentanil
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Remi 0.1 (Experimental): Following intravenous (IV) administration of 0.5 mg Atropine (Atropin, Biofarma, Istanbul, Turkey) prior to the induction, the patients randomly (by lot) received one of the three different doses [(0.1), 0.2, 0.3 µg/kg/min] of remifentanil infusion (Ultiva, Glaxo Wellcome, Marly-le-Roi, France) for two minutes.
  Interventions: Drug: Remi 0.1
- Remi 0.2 (Experimental): Following intravenous (IV) administration of 0.5 mg Atropine (Atropin, Biofarma, Istanbul, Turkey) prior to the induction, the patients randomly (by lot) received one of the three different doses [0.1, (0.2), 0.3 µg/kg/min] of remifentanil infusion (Ultiva, Glaxo Wellcome, Marly-le-RoiFrance) for two minutes.
  Interventions: Drug: Remi 0.2
- Remi 0.3 (Experimental): Following intravenous (IV) administration of 0.5 mg Atropine (Atropin, Biofarma, Istanbul, Turkey) prior to the induction, the patients randomly (by lot) received one of the three different doses [0.1, 0.2, (0.3) µg/kg/min] of remifentanil infusion (Ultiva, Glaxo Wellcome, Marly-le-Roi, France) for two minutes.
  Interventions: Drug: Remi 0.3

INTERVENTIONS:
Drug: Remi 0.1 — Intravenous (IV) administration of 0.5 mg Atropine prior to the induction, the patients randomly (by lot) received one of the three different doses (0.1 µg/kg/min) of remifentanil infusion for two minutes.After 2-minute remifentanil infusion, 0.5 mg/kg propofol was administered via IV route increasing the dose by 10 mg every 10 seconds; 0.5 mg/kg rocuronium was administered via IV route at the time of loss of eyelash reflex and consciousness. Two minutes later, intubation was performed. After recording the baseline values of heart rate, systolic arterial pressure, mean arterial pressure and diastolic arterial pressure, which were planned to be investigated, and administering atropine, a total of six measurements at one-minute intervals were performed until the time of intubation.
  Other Names: remifentanil, Ultiva, Glaxo Wellcome, Marly-le-Roi, France
  Arms: Remi 0.1
Drug: Remi 0.2 — .Intravenous (IV) administration of 0.5 mg Atropine prior to the induction, the patients randomly (by lot) received one of the three different doses (0.2 µg/kg/min) of remifentanil infusion for two minutes.After 2-minute remifentanil infusion, 0.5 mg/kg propofol was administered via IV route increasing the dose by 10 mg every 10 seconds; 0.5 mg/kg rocuronium was administered via IV route at the time of loss of eyelash reflex and consciousness. Two minutes later, intubation was performed. After recording the baseline values of heart rate, systolic arterial pressure, mean arterial pressure and diastolic arterial pressure, which were planned to be investigated, and administering atropine, a total of six measurements at one-minute intervals were performed until the time of intubation.
  Other Names: remifentanil, Ultiva, Glaxo Wellcome, Marly-le-Roi, France
  Arms: Remi 0.2
Drug: Remi 0.3 — Intravenous (IV) administration of 0.5 mg Atropine prior to the induction, the patients randomly (by lot) received one of the three different doses (0.3 µg/kg/min) of remifentanil infusion for two minutes.After 2-minute remifentanil infusion, 0.5 mg/kg propofol was administered via IV route increasing the dose by 10 mg every 10 seconds; 0.5 mg/kg rocuronium was administered via IV route at the time of loss of eyelash reflex and consciousness. Two minutes later, intubation was performed. After recording the baseline values of heart rate, systolic arterial pressure, mean arterial pressure and diastolic arterial pressure, which were planned to be investigated, and administering atropine, a total of six measurements at one-minute intervals were performed until the time of intubation.
  Other Names: remifentanil, Ultiva, Glaxo Wellcome, Marly-le-Roi,
  Arms: Remi 0.3

SUMMARY:
Effects of different doses of remifentanil on hemodynamic response to anesthesia induction in elderly patients ABSTRACT OBJECTİVE: The investigators compared the effects of three different doses of remifentanil infusion, which have been performed for the induction of anesthesia in elder patients, on cardiovascular response.

PATIENTS AND METHODS: The present study was designed as a randomized, prospective and double-blind study. A total of 90 ASA I-II patients over the age of 65 years were enrolled and each group consisted of 30 subjects. The patients were randomly (by lot) assigned to receive one of the three doses of remifentanil infusion (0.1, 0.2 or 0.3 µg/kg/min) for two minutes. Subsequently, 0.5 mg/kg propofol was administered via IV route and, 0.5 mg/kg rocuronium was administered via IV route at the time eyelash reflex disappeared. Intubation was performed after two minutes. After recording baseline values of heart rate (HR), systolic arterial pressure (SBP), diastolic arterial pressure (DBP) and mean arterial pressure (MAP), these values were recorded at the 1st, 2nd, 3rd, 4th and 5th minutes of induction.

DETAILED DESCRIPTION:
The present study was carried out after the approval of "Dokuz Eylül University School of Medicine, Clinical Researches Ethics Committee and informed consents of the patients were obtained. A total of 90 normotensive and American Society of Anesthesiology (ASA) I-II patients at and over the age of 65 years undergoing elective non-cardiac surgery were enrolled in the study. The study was designed as a prospective, randomized, double-blind study. The patients were randomly (sealed envelope method) assigned to one of the following groups:

Remi 0.1= dose of remifentanil for the induction of anesthesia is 0.1 µg/kg/min (n=30) Remi 0.2= dose of remifentanil for the induction of anesthesia is 0.2 µg/kg/min (n=30) Remi 0.3= dose of remifentanil for the induction of anesthesia is 0.3 µg/kg/min (n=30) The patients and the anesthesiologist, who would perform the induction of anesthesia, were blind for remifentanil dose.

In all patients, an intravenous (IV) line was opened on the dorsum of the left hand using 18-Gauge cannula before they were admitted to the surgery room and 0.9% isotonic NaCl solution was infused at a dose of 5-7 mL/kg without any agent for premedication. The patients underwent standard monitoring composed of electrocardiogram (ECG), pulse oximeter, noninvasive blood pressure measurement, and end tidal carbon dioxide measurement. After 5-minute stabilization period following monitoring, heart rates and systemic arterial pressures of the patients were measured and baseline values were recorded for each patient (6). Measurement of systemic arterial pressure was done by automatic oscillometry (Hewlett-Packard HP M1008B) and heart rate (HR) was calculated on the ECG trace (Hewlett-Packard HP M1002A). Induction of Anesthesia Following routine monitoring in the surgery room, induction of anesthesia was started after the patients were peroxygenized and received 0.9% isotonic NaCl solution via IV route at a dose of 5-7 mL/kg. Following intravenous (IV) administration of 0.5 mg Atropine (Atropin, Biofarma, Istanbul, Turkey) prior to the induction, the patients randomly (by lot) received one of the three different doses (0.1, 0.2, 0.3 µg/kg/min) of remifentanil infusion (Ultiva, Glaxo Wellcome, Marly-le-Roi, France) for two minutes. After 2-minute remifentanil infusion (remi concentration of 40 µg/mL), 0.5 mg/kg propofol ( Propofol 1% Fresenius; Fresenius Kabi, Uppsala, Sweden) was administered via IV route increasing the dose by 10 mg every 10 seconds; 0.5 mg/kg rocuronium was administered via IV route at the time of loss of eyelash reflex and consciousness (7). Two minutes later, intubation was performed at one sitting in all patients by a specialist with at least 5-year experience using Macintosh laryngoscope. The lungs were manually ventilated by sevoflurane at an inspiratory concentration of 1.5% and by 50% air/oxygen until the intubation. Infusion dose of remifentanil, which had been performed at induction dose until intubation, was decreased by 50% in all groups after intubation.

The maintenance of anesthesia was provided with remifentanil at predetermined dose and the ventilation continued with 50% air/oxygen and sevoflurane at an inspiratory concentration of 1.5% in the way target end-tidal carbon dioxide value would be 30-35 mmHg.

After recording the baseline values of heart rate, systolic arterial pressure, mean arterial pressure and diastolic arterial pressure, which were planned to be investigated, and administering atropine, a total of six measurements at one-minute intervals were performed until the time of intubation; no measurement was performed during intubation period.

Hypotension was defined as a systolic arterial pressure < 90 mmHg or a decrease more than 30% of the baseline value, and it was treated with 5 mg IV Ephedrine (Efedrin, Osel, Istanbul, Turkey) (8). Determining 40% or higher decrease in the above-mentioned values, the dose of remifentanil infusion was decreased by 50% in addition to administration of 5 mg IV Ephedrine; in case no improvement was observed and systolic arterial pressure remained below 40% of the baseline value, the dose of remifentanil was decreased by 1/4. A heart rate < 50/min was defined as bradycardia and treated with 0.5 mg IV Atropine.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive patients
* ASA I-II
* Patients over the age of 65 years
* Undergoing elective non-cardiac surgery

Exclusion Criteria:

* Patients who had allergy against opioids
* Chronic benzodiazepine, opioid, alcohol or substance users
* Obese (body mass index > 30)
* Expected to have difficult airway
* Patients had hypertension
* Patients have been receiving any drug influencing the cardiovascular system (beta -adrenergic blocker, calcium channel blocker, etc.)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Measurement was performed using physiological parameters. After recording baseline values of systolic arterial pressure (SBP), these values were recorded at the 1st, 2nd, 3rd, 4th and 5th minutes of induction. | Five minutes
  Aim to identify the remifentanil dose that we can recommend. To determine hemodynamic changes likely to occur while using three different doses of remifentanil in the induction of anesthesia in the patients at and over the age of 65 years. Physiological parameters; measurement of systemic arterial pressure was done by automatic oscillometry (Hewlett-Packard HP M1008B).
Measurement was performed using physiological parameters. After recording baseline values of diastolic arterial pressure (DBP), these values were recorded at the 1st, 2nd, 3rd, 4th and 5th minutes of induction. | Five minutes
  Aim to identify the remifentanil dose that we can recommend. To determine hemodynamic changes likely to occur while using three different doses of remifentanil in the induction of anesthesia in the patients at and over the age of 65 years. Physiological parameters; measurement of diastolic arterial pressure was done by automatic oscillometry (Hewlett-Packard HP M1008B).
Measurement was performed using physiological parameters. After recording baseline values of mean arterial pressure (MBP), these values were recorded at the 1st, 2nd, 3rd, 4th and 5th minutes of induction. | Five minutes
  Aim to identify the remifentanil dose that we can recommend. To determine hemodynamic changes likely to occur while using three different doses of remifentanil in the induction of anesthesia in the patients at and over the age of 65 years. Physiological parameters; measurement of mean arterial pressure was done by automatic oscillometry (Hewlett-Packard HP M1008B).
Measurement was performed using physiological parameters. After recording baseline values of heart rate (HR), these values were recorded at the 1st, 2nd, 3rd, 4th and 5th minutes of induction. | Five minutes
  Aim to identify the remifentanil dose that we can recommend. To determine hemodynamic changes likely to occur while using three different doses of remifentanil in the induction of anesthesia in the patients at and over the age of 65 years. Physiological parameters; measurement of heart rate was calculated on the ECG trace (Hewlett-Packard HP M1002A).

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Boztas, MD, Principal Investigator — Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation Inciraltı IZMIR 35320

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Boztas N, Oztekin S, Ozkardesler S, Akan M, Ozbilgin S, Baytok A. Effects of different doses of remifentanil on hemodynamic response to anesthesia induction in healthy elderly patients. Curr Med Res Opin. 2017 Jan;33(1):85-90. doi: 10.1080/03007995.2016.1239189. Epub 2016 Oct 17. PMID 27646937